CLINICAL TRIAL: NCT04766268
Title: Prostate Artery Embolizaton: Single Center Experience
Brief Title: Prostate Artery Embolization: Single Center Experience
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Jay Vasani, Assistant Professor, University of Mississippi Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020V0337
Record Dates: First submitted 2021-01-11; First posted 2021-02-23 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2021-02

CONDITIONS: Benign Prostatic Hyperplasia (BPH); Lower Urinary Tract Symptoms
Keywords: PAE; Prostate artery embolization; Prostatic artery embolization; BPH; Lower urinary tract symptoms
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Intervention Model Description: Prospective, single arm
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PAE group (Experimental): Patients with BPH with moderate lower urinary tract symptoms fulfilling the inclusion criteria and exclusion criteria will be enrolled in the trial to determine safety and effectiveness of prostate artery embolization and determine factors associated with improved procedure outcome.
  Interventions: Other: Prostate artery embolization

INTERVENTIONS:
Other: Prostate artery embolization — Prostate artery embolization (PAE) is a safe and effective minimally invasive interventional radiology procedure in which intraprostatic vessels are embolized to shrink the size of the prostate gland. LUTS is mainly categorized into irritative, obstructive, and mixed types. This has a variable impact on patients' quality of life by interfering with sleep, activities of daily living, anxiety, mobility, leisure, and effect on sexual activities. This trial aims to determine safety and effectiveness of prostate artery embolization and determine factors associated with improved procedure outcome.
  Other Names: PAE

SUMMARY:
Benign prostatic hyperplasia (BPH) is an enlarged prostate gland from smooth muscle and glandular hyperplasia seen in the aging population with a prevalence of upto 90% in patients in the ninth decade. Lower urinary tract symptoms (LUTS) and bladder outlet obstruction (BOO) are the most common presenting symptoms of BPH. Patients are initially evaluated with a complete history and physical exam to rule out other causes of LUTS and assess the severity of LUTS with scoring systems such as the American Urologic Association Symptom Index (AUASI) or the International Prostate Symptom Score (IPSS). Patients with mild or no symptoms are treated with watchful waiting. Surgical procedure such as transurethral resection of the prostate and minimally invasive procedures such as microwave ablation and prostate artery embolization are performed in patients with failed medical management or patients who are not able to tolerate the side effects of the medications. Prostate artery embolization is a safe minimally invasive procedure shown to improve IPSS and quality of life with none or potential risk of minor complications shown in short, intermediate, and long term follow up.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is an enlarged prostate from smooth muscle and glandular hyperplasia that results in lower urinary tract symptoms due to bladder outlet obstruction. It is seen in 8% of men in the fourth decade with increased prevalence to up to 90% of men in the ninth decade (1). Patients typically present with groups of symptoms referred to as lower urinary tract symptoms (LUTS) of which may include urgency, frequency, nocturia, incomplete bladder emptying, and weak urinary stream (2). LUTS is mainly categorized into irritative, obstructive, and mixed types. This has a variable impact on patients' quality of life by interfering with sleep, activities of daily living, anxiety, mobility, leisure, and effect on sexual activities (3). The risk factors for developing BPH include African American race, obesity, type 2 diabetes mellitus, high levels of alcohol consumption, and physical inactivity (4).

Patients with LUTs are evaluated with a complete history and physical to rule out causes other than BPH and bladder dysfunction such as excess fluid and caffeine intake, and use of medications including diuretics and antihistamine. Patients are further evaluated with screening tools such as the American Urologic Association Symptom Index (AUASI) or the International Prostate Symptom Score (IPSS) to determine the severity of LUTS secondary to BPH. IPSS is an 8 question screening tool that assesses the quality of life in addition to 7 questions in AUASI (4). Each question is scored from 0 to 5 and a minimum change of 3 points is considered a clinically important difference (5). Patients with AUASI score of less than 8 are considered to have mild or no symptoms and are managed with watchful waiting (6). Moderate or severe symptoms are considered in patients with AUASI score of 8 or greater than 8 and are managed with pharmacologic treatment including alpha-adrenergic receptor blockers, 5 alpha-reductase inhibitors, antimuscarinic agents, and phosphodiesterase 5 inhibitors. Additionally, international index of erectile function (IIEF) is used to further assess quality of life. For patients who have failed medical management, experience side effects from medications, or not interested in medical therapy are offered minimally invasive surgical treatment such as microwave ablation, surgical treatment including open prostatectomy and transurethral resection of the prostate (TURP) and interventional radiology procedure, prostate artery embolization.

Prostate artery embolization (PAE) is a safe and effective minimally invasive interventional radiology procedure in which intraprostatic vessels are embolized to shrink the size of the prostate gland. Preprocedural assessment includes IPSS, the international index of erectile function (IIEF-5) to asses pre-existing erectile dysfunction (7), postvoid residual (PVR) to objectively assess the degree of bladder outlet obstruction, cross-sectional imaging of the prostate gland, and screening for prostate cancer (8). The current indication for PAE is patients with moderate or severe LUTS from BPH who have not responded to medications or find medication side effects to be intolerable. Patients are excluded from the procedure in other causes of LUTS such as prostate cancer, neurogenic bladder prostatitis, urethral strictures. Clinical trials are underway that demonstrate the efficacy of the procedure and define indications and contraindications. Meta-analysis showed a statistically significant decrease in IPSS of 12.9, 15, 15, and 20.4 points from baseline at 1, 3, 6, 12 months, respectively (9). Additionally, statistically significant improvement in the quality of life and PVR were noted at 1, 3, 6, 12 months. An overall incidence of a compilation was 32.9% (9), the majority of which were classified as minor per SIR guidelines. Rectalgia, dysuria, and transient urinary retention were the most frequent minor complications of PAE. A few major complications related to PAE were severe urinary tract infection and bladder ischemia

ELIGIBILITY:
Inclusion Criteria:

* Anyone with international prostate symptom score greater than or equal to 8 (moderate to severe lower urinary tract symptoms)
* Quality of life assessment greater than 3
* Prostate volume greater than 40 cm3
* Men >45 years old
* Indwelling urinary catheter secondary to benign prostatic hyperplasia or moderate-severe lower urinary tract symptoms

Exclusion Criteria:

* Evidence of tortuous or severe atherosclerotic vessels on CT
* Neurogenic bladder
* <8 international prostate symptoms score
* Prostate volume less than 40cm3
* History of prostate cancer

Min Age: 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-04-10 (Estimated)

PRIMARY OUTCOMES:
Change in international prostate symptom score from baseline | Baseline, 1 month, 3 months, 6 months, 1 year and 2 years
  IPSS is an assessment of patient's lower urinary tract symptoms which categorizes the symptoms into Mild (1-7), Moderate (8-19) Severe (20-35). Decrease in the score means favorable outcome. This score will measured during each follow up visit.
Change in quality of life assessment from baseline | Baseline, 1 month, 3 months, 6 months, 1 year and 2 years
  Improvement of QOL from baseline. Scores include 0 - Delighted, 1- Pleased, 2- Mostly satisfied, 3 - Mixed, 4- mostly dissatisfied, 5 - Unhappy and 6 - Terrible
Change in post-void residual volume from baseline | Baseline, 1 month, 3 months, 6 months, 1 year and 2 years
  Improvement of PVR (Post void residue) compared to baseline. This will be performed with either an US or automated bladder scanner demonstrating volume of urine remaining in the urinary bladder after urination.
Successful removal of foley catheter in patient | Baseline, 1 month, 3 months, 6 months, 1 year and 2 years
  This outcome will be assessed for only those patients who are already wearing a foley catheter due to BPH related obstruction. Number of these patients cannot be predetermined. These patients will undergo the procedure while they are wearing the catheter. Once the procedure is performed they will return to the clinic for voiding trial (assess if the foley can be removed).Success in removal of foley catheter after spontaneous voiding with PVR <200 ml. Favorable outcome will be that the patient is able to void freely without needing a foley catheter.

SECONDARY OUTCOMES:
Change in prostate volume | Baseline, 3 months
  Reduction in prostate volume at 3 months measured by US or MRI
Change in international index of erectile function | Baseline, 1 month, 3 months, 6 months, 1 year and 2 years
  Change in IIEF/SHIM score compared to baseline. This score is a measure of severity of erectile dysfunction where score of 22-25 (No ED), 17-21 (mild ED), 12-16 ( mild to moderate), 8-11 (moderate), 5-7 (Severe)
Determine the need for medication use after PAE | 1 month, 3 months, 6 months, 1 year and 2 years
  To determine successful cessation of BPH medicines at 1month post PAE

CONTACTS AND LOCATIONS:
Overall Officials: Jay Vasani, MD, Principal Investigator — University of Mississippi Medical Center; Chadwick Huckabay, MD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical center, Jackson, Mississippi, United States